CLINICAL TRIAL: NCT03888118
Title: Clinical Efficacy of Luna EMG Robot Therapy for Patients After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rehamed Center (Other)
Responsible Party: Principal Investigator, Marzena Adamczyk, Investigator, Rehamed Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2019-03-19; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Stroke
Keywords: Luna EMG; drop foot; chronic stroke
MeSH Terms: conditions — Stroke; Peroneal Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): A four-week rehabilitation program (Monday to Friday) involving the hour of individual ankle therapy and one hour therapy on the Luna EMG device.
  Interventions: Device: Luna EMG
- Control group (No Intervention): A four-week rehabilitation program (Monday to Friday) involving two hours of individual ankle therapy.

INTERVENTIONS:
Device: Luna EMG — The duration of the overall therapeutic intervention in both groups will be the same.
  Arms: Study Group

SUMMARY:
A lot of studies prove that rehabilitation with the use of modern devices accelerates the recovery of function in patients after stroke. Repeated correct movement patterns affect the central nervous system and stimulating its plasticity. Despite the fact that so many studies confirm the validity of therapy using robots, it is still difficult to assess to what extent its use improves the effectiveness of traditional therapy. In these studies, we want to objectively assess the effectiveness of the Luna device using EMG biofeedback.

ELIGIBILITY:
Inclusion Criteria:

* patients over 6 months after stroke,
* tibialis anterior strength (Lovett scale) not less than 1 and not greater than 3,
* Ashworth scale in tibialis anterior 0,1, 2

Exclusion Criteria:

* patients less than 6 months after stroke,
* tibialis anterior strength (Lovett scale) 0, 4, 5,
* Ashworth scale in tibialis anterior higher than 2,
* damage to the central nervous system which is another incident,
* serious cognitive deficit,
* stiffness of the ankle.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
EMG using the Luna EMG | 3 minutes
  EMG will be performed using the Luna EMG device also allowing the treatment and diagnosis. With Luna EMG we can supply objective, data driven diagnosis. Innervation diagnosis and motor unit recruitment through surface electromyography. We'd like to assess bioelectrical activity at the tibialis anterior muscle during relaxing for two minutes (mean, minimum and maximum electrical activity in muscle - in microvolts).
EMG using the Luna EMG | 1 minute
  EMG will be performed using the Luna EMG device also allowing the treatment and diagnosis. With Luna EMG we can supply objective, data driven diagnosis. Innervation diagnosis and motor unit recruitment through surface electromyography. We'd like to assess bioelectrical activity at the tibialis anterior muscle activation patterns during three times dorsiflexion (mean, minimum and maximum electrical activity in muscle - in microvolts).
Lovett scale | 1 minute
  The muscle strength in Lovett scale is graded on a scale of 0-5:
  Grade 5: Muscle contracts normally against full resistance. Grade 4: Muscle strength is reduced but muscle contraction can still move joint against resistance.
  Grade 3:Muscle strength is further reduced such that the joint can be moved only against gravity with the examiner's resistance completely removed.
  Grade 2: Muscle can move only if the resistance of gravity is removed. Grade 1: Only a trace or flicker of movement is seen or felt in the muscle or fasciculations are observed in the muscle.
  Grade 0: No movement is observed. Higher values represent a better outcome. We'd like to asses foot dorsiflexor muscle strength.
Ashworth scale | 1 minute
  Measurement of resistance during passive plantarflexion and dorsiflexion.
  Scorse range from 0 to 4, with 5 choices:
  Grade 0: No increase in muscle tone. Grade 1: Slight increase in muscle tone, manifested by a catch and release or by minimal.
  resistance when the affected part is moved in flexion or extension. Grade 2: More marked increase in muscle tone, but affected part(s) easily moved.
  Grade 3: Considerable increase in muscle tone, passive movement difficult. Grade 4: Affected part(s) rigid in flexion or extension. Higher values represent a worse outcome.
Tinetti test - gait and balance | 10 minutes
  The Tinetti Balance and Gait test is a standardized evaluation of mobility and stability. Balance and gait are assessed and scored individually in a 16-item test. A three-point ordinal scale, ranging from 0-2. "0" indicates the highest level of impairment and "2" the individuals independence. Gait is scored 0-12 and balance is scored 0-16. Total Test Score is maximum 28.
  Interpretation:
  25-28 low fall risk 19-24 medium fall risk < 19 high fall risk Higher score represent a better outcome.